CLINICAL TRIAL: NCT03965650
Title: Randomized Controlled Study of a Video Coaching Program of Physical Activity in Patients Suffering From Axial Spondyloarthritis
Brief Title: Video Coaching of Physical Activity in Axial Spondyloarthritis
Acronym: SatiSpAction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP190622; 2019-A01384-53 (Registry Identifier: IDRCB)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Axial Spondyloarthritis
Keywords: axial spondyloarthritis; online video coaching; physical activity
MeSH Terms: conditions — Axial Spondyloarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: video coaching exercises (Experimental): Video coaching exercises group: patients will perform physical exercises according to a video coaching program 3 times weekly during 6 months. The on-line program has been designed especially for this study.
  Interventions: Other: Video coaching exercises
- Control group: routine exercises (Active Comparator): Routine method advising and encouraging patients to perform physical activities according to the WHO recommendations during 3 months then to follow the video coaching physical exercises program during 3 months.
  Interventions: Other: Routine exercises

INTERVENTIONS:
Other: Video coaching exercises — Patients will perform physical exercises following a specifical video coaching program during 6 months.
  Arms: Intervention group: video coaching exercises
Other: Routine exercises — Routine method by advising and encouraging patients to perform exercises according to the WHO recommendations during the first 3 months of the study.
  Thereafter, patients will have access to the video coaching program of physical activities during the following 3 months.
  Arms: Control group: routine exercises

SUMMARY:
The primary objective of the study is to demonstrate the beneficial effect of a 3 months home-based physical exercise program supervised by online videos, in addition to the usual recommendations, in comparison with usual physical activity as recommended by the WHO.

The secondary objectives of the study are :

1. to compare the following criteria between 2 groups at 3 and 6 months:

   * quality of life;
   * other measures of disease activity ;
   * sleep quality ;
   * walking ability
   * muscle strength of;
   * professional activity;
   * cost of cares;
   * evolution of weight, BMI and waist.
2. to evaluate the observance of physical activity program and its tolerance at 3 and 6 months.

DETAILED DESCRIPTION:
The spondyloarthritides are a group of inflammatory rheumatic diseases, including ankylosing spondylitis, reactive arthritis, inflammatory bowel disease-related rheumatic disease, and psoriatic arthritis.

The frequence of axial spondyloarthritis is 0.41% in the french population. This disease is associated with a reduction of physical capacities and quality of life. NSAIDs or even biologic therapies do not always permit a sufficient control of the disease. Different physical exercise programs can be effective as an additional therapy for spondyloarthritis, with positive effects on spinal mobility as well as main disease activity and functional indices (BASDAI, BASFI and BASMI). The severity of the disease does not seem to influence significantly the patients' motivation in practicing physical activity.

This proposed study aims to demonstrate the beneficial effect of physical exercises coached with a specific internet program diffused on a secured platform.

Each patient will have to connect 3 times weekly in order to follow the entire program.

The impact will be evaluated at 3 months and 6 months.

Potential impacts of video-coaching program are:

* reduction of the intrinsic inflammatory activity of the rheumatic disease;
* improvement of the global physical condition: muscular strength and resistance, walking ability, chest expansion;
* reduction of fatigue and improvement of sleeping;
* reduction of consumption of symptomatic drug (analgesics, NSAIDs, corticosteroids).

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 65 years;
* Patient can read and understand French;
* Signed informed consent form to participate in the study;
* Axial spondylarthritis according to ASAS criteria;
* Patient with a BASDAI score between 2.5 and 5;
* No change of biotherapy anti-TNF or anti-IL17 during the 3 months preceding the inclusion;
* Patient equipped with an internet access;
* Medical certificate of proposed physical activities.

Exclusion Criteria:

* All diseases (cardiovascular disease or chronic neurological disease or others) contraindicating the requested exercises according to physician;
* Axial spondyloarthritis in remission defined by a BASDAI < 2.5/10 or in excessive inflammatory activity, defined by BASDAI > 5/10;
* Pregnant woman (positive pregnant test) or woman try to conceive in following 6 months;
* Patient with articular prosthesis;
* Patient who already participate in a specific exercise program or practice a sport (including Yoga or Tai Chi) more than one hour per week;
* Severe obesity ( BMI > 35);
* Patient without health insurance;
* Patient legally unable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients responding to the "ASAS 20" criterion at 3 months | at 3 months
  The primary outcome measure will be the proportion of patients simultaneously satisfying both criteria :
  * at least 20% improvement
  * improvement of at least 10 points on visual analog scale in the following domains: overall evaluation by the patient, visual analog scale (pain scale), Bath Ankylosing Spondylitis Functional Index (BASFI), and Bath Ankylosing Spondylitis Disease Activity Index (BASDAI).

SECONDARY OUTCOMES:
Ankylosing Spondylitis Disease Activity : (BASDAI) (PRO) | at baseline, 3 months and 6 months
  Ankylosing Spondylitis Disease Activity will be assessed with the Bath Ankylosing Spondylitis Disease Activity (BASDAI) auto-questionnaire assessing the inflammatory activity of the disease.
Ankylosing Spondylitis Disease Activity : (ASDAS CRP) (PRO) | at baseline, 3 months and 6 months
  Ankylosing Spondylitis Disease Activity will be assessed with the Ankylosing Spondylitis Disease Activity Score (ASDAS CRP) auto-questionnaire assessing the inflammatory activity of the disease.
Bath Ankylosing Spondylitis Functional Index (BASFI) (PRO) | at baseline, 3 months and 6 months
  Data collected with the Bath Ankylosing Spondylitis Functional Index (BASFI) auto-questionnaire assessing the functional impact of disease.
Fatigue (PRO) | at baseline, 3 months and 6 months
  Fatigue will be assessed with a Visual Analogue Scale
Health assessment: HAQ-S (PRO) | at baseline, 3 months and 6 months
  SpA-related health will be assessed with the Health Assessment Questionnaire for the Spondyloarthropathies (HAQ-S)
SPA impact on general health: ASAS-HI (PRO) | at baseline, 3 months and 6 months
  General health will be assessed with the ASAS Health Index auto-questionnaire
Work Productivity and Activity : WPAI (PRO) | at baseline, 3 months and 6 months
  Work Productivity and Activity will be assessed with the Work Productivity and Activity Impairment (WPAI) auto-questionnaire
Sleep quality: PSQI | at baseline, 3 months and 6 months
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI) auto-questionnaire
Physical activity: IPAQ (PRO) | at baseline, 3 months and 6 months
  Physical activity will be assessed with the International Physical Activity Questionnaire (IPAQ) - Short Form and Long Form auto-questionnaires
Analgesic and anti-inflammatory drug intake | at 3 months and 6 months
  Following drugs intake will be collected:
  * non-steroidal anti-inflammatory drugs (NSAIDs)
  * corticosteroids
Anthropometric measures: BASMI | at baseline, 3 months and 6 months
  The functional impact of SpA will be assessed with the Bath Ankylosing Spondylitis Metrology Index (BASMI)
Anthropometric measures: Enthesitis: MASES | at baseline, 3 months and 6 months
  Entesis involvement will be assessed with the Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Anthropometric measures: Muscle strength: dynamometer | at baseline, 3 months and 6 months
  Muscle strength of the upper and lower limbs will be assessed with a dynamometer
Anthropometric measures: 6-minutes walk test | at baseline, 3 months and 6 months
  Walking ability will be assessed with the 6-minutes walking test.
Anthropometric measures: Body mass index (BMI) | at baseline, 3 months and 6 months
  Weight, height and waist size will be collected to calculate the BMI of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Le Goux, MD, Principal Investigator — Service de rhumatologie, Hôpital Ambroise Paré; Gilles Hayem, MD, Study Director — Service de rhumatologie, Hôpital Saint Joseph, 185 Rue Raymond Losserand 75014 Paris
Locations (1):
- Service de rhumatologie, Hôpital Ambroise Paré, Boulogne-Billancourt, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No